CLINICAL TRIAL: NCT02111655
Title: Second Generation Surveillance Techniques to Prevent Thrombosis and Increase Assisted Primary Patency in Native Arteriovenous Fistula. A Prospective Controlled Trial.
Brief Title: Improving Arteriovenous Fistula Patency
Acronym: METTRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Infanta Sofia (Other)
Responsible Party: Principal Investigator, Antonio Cirugeda, Principal Investigator, Hospital Infanta Sofia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 210443-031132-261233; 3598 (Other: CEIC HOSPITAL UNIVERSITARIO DE LA PAZ)
Record Dates: First submitted 2014-03-28; First posted 2014-04-11 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Thrombosis
Keywords: Thrombosis; Arteriovenous fistulae; Hemodialysis; Doppler ultrasound; Vascular access blood flow; Surveillance
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clasical Surveillance of AVF (Other): Classical evaluation of AVF includes:
  1. Vital sings and predialysis physical examination of AVF every dialysis session.
  2. Effective blood flow, venous pressure, arterial pressure, at the beginning and at the end of the dialysis session.
  3. Weekly ktv test using biosensors or monthly if using monocompartimental Daugirdas equation.
  4. Quarterly recirculation with urea method.
  Following Spanish Nephrology VA guidelines will be consider as alarm criteria:
  1.25% Increased venous pressure. 2.25% Decreased pump blood flow. 3.0,2 ktv decreased compared with previous measurement. 4.> 10% recirculation using urea method. 5.Prolonged coagulation time or cannulation difficulties in 3 consecutive dialysis sessions.
  6.Pathologic physical examination with any other criteria.
  Interventions: Procedure: vital signs; Procedure: physical examination of AVF; Procedure: ktv test; Procedure: urea method
- Second generation surveillance of AVF (Experimental): In addition to the classical surveillance and monitoring methods, in the experimental group Doppler ultrasound and transonic dilution method will be performed on a quarterly basis.
  In addition to the classical alarm criteria and derived from the results in Doppler ultrasound an transonic dilution method the following alarm criteria would also be considered in the experimental group:
  1. 25% or higher decreased in QA compared with previous measurement.
  2. QA lower than 500 ml/min.
  3. Stenotic area with a higher than 50% reduction of blood vessel lumen would be considered as alarm criteria only if it comes with a haemodynamic repercussion criteria defined as Peak systolic velocity (PSV) higher than 400 cm/sc, aliasing, or PSV ratio stenosis/pre-stenosis higher than 3.
  Interventions: Device: Second generation surveillance of AVF; Procedure: vital signs; Procedure: physical examination of AVF; Procedure: ktv test; Procedure: urea method

INTERVENTIONS:
Device: Second generation surveillance of AVF — Doppler ultrasound and transonic dilution method technique will be performed in the experimental group quarterly.
  QA will be measured by both techniques and haemodynamic repercussion stenosis will be evaluated by doppler ultrasound.
  Other Names: Doppler ultrasound: M-Turbo. Sonosite.; Transonic dilution method: Transonic System Inc HD-03
  Arms: Second generation surveillance of AVF
Procedure: vital signs — Effective blood flow, venous pressure, arterial pressure, at the beginning and at the end of the dialysis session
Procedure: physical examination of AVF — Predialysis physical examination of AVF every dialysis session.
Procedure: ktv test — Weekly ktv measurement using biosensors. In patients who have been dialyzed in monitors with no biosensors, ktv will be measured monthly using monocompartimental Daugirdas equation
Procedure: urea method — Quarterly recirculation with urea method.

SUMMARY:
All vascular access guidelines recommend monitoring and surveillance protocols to prevent vascular access complications in hemodialysis units.

However, in the case of second generation screening techniques which determine access blood flow measurement (QA), there is a huge controversy about it´s efficiency.

Although multiple observational studies find a decrease in the thrombosis rate and an increased primary assisted patency survival related to the use of these techniques, a recently published meta-analysis find contradictory results in the randomized controlled trials, affirming that the measurement of QA is useless in grafts and questionable in native arteriovenous fistulae (AVF).

We have designed a multicenter, prospective, open label, controlled, randomized trial, to prove the usefulness of the QA measurement using two complementary second generation techniques, Doppler ultrasound and Transonic dilution method, compared to the classical monitoring and surveillance methods.

The primary endpoint will be a reduction in the thrombosis rate with an increased assisted primary patency survival, and a cost effectiveness economic analysis.

As secondary endpoints we will analyze the impact over non-assisted primary patency survival and secondary patency survival.

DETAILED DESCRIPTION:
Definition:

Multicenter, prospective, open label, controlled, randomized trial, to prove the usefulness of the QA measurement using two complementary second generation techniques, Doppler ultrasound and Transonic dilution method, compared to the classical monitoring and surveillance methods.

For Patient Registries:

Clinical data repository (CDR) paper notebook will contain all baseline patient characteristics and the information related to vascular access. These data will be collected by the different investigators and reviewed and included in data base by the study´s monitor.

This information will be included in a centralized computer database (SPSS 15.0 computer system) and encoded in order to preserve patients´ confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signature.
* Age between 18 and 95 years old.
* Functioning native AVF.
* Patients with end stage renal disease (ESRD) undergoing hemodialysis program for at least three months.

Exclusion Criteria:

* Coagulopathy or hemoglobinopathy of any cause.
* Hospitalization of any cause in the previous month.
* VA related complications or dysfunction in the previous three months.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2012-09-01; Primary Completion 2015-09-29 (Actual); Study Completion 2015-09-29 (Actual)

PRIMARY OUTCOMES:
Improved primary patency rate in arteriovenous fistulae with the use of doppler ultrasound and transonic dilution method | Up to 3 years follow up
  Differences in assisted primary patency rates (thrombosis free access survival) in AVF between the two groups: control group in which classical monitoring and surveillance techniques are applied and experimental group in which Doppler ultrasound and transonic were performed every three months in addition to classical methods.
  Cost efficacy analysis in both groups will be done, measuring all vascular access (VA) related health care spending (VA hospitalization costs, central venous catheter (CVC) placements, surgeries and endovascular procedures will be recorded).

SECONDARY OUTCOMES:
Compared non-assisted primary patency rates (intervention free access survival) and secondary patency rates (access survival until abandonment) between the two groups. | Up to 1 year follow up
Evaluate the efficacy and efficiency of second generation methods | Up to 2 years follow up
  It will be evaluated the positive and negative predictive value of each second generation technique, doppler ultrasound and Transonic dilution method. The accuracy of these techniques will be compared to determine which one show more benefits detecting pathology of AVF.
Reproducibility in Doppler ultrasound technique | Up to 3 years follow up.
  There will be always two observers for each doppler ultrasound (same observers for same AVF). Differences among different quarterly measures in stable AVF will be evaluated, as well as the differences between the two observers in QA measurement.
Possible influence of different baseline items in the risk of thrombosis of native AVF | Up to 3 years follow up
  It will be evaluated if there is any influence of age, body mass index, use of antiplatelet therapy, anticoagulant therapy or the use of pentoxifylline in the risk of thrombosis of AVF
Compared non-assisted primary patency rates (intervention free access survival) and secondary patency rates (access survival until abandonment) between the two groups. | Up to 2 years follow up
Evaluate the efficacy and efficiency of second generation methods | Up to 3 years follow up
  It will be evaluated the positive and negative predictive value of each second generation technique, doppler ultrasound and Transonic dilution method. The accuracy of these techniques will be compared to determine which one show more benefits detecting pathology of AVF.
Compared non-assisted primary patency rates (intervention free access survival) and secondary patency rates (access survival until abandonment) between the two groups. | Up to 3 years follow up

CONTACTS AND LOCATIONS:
Overall Officials: ANTONIO CIRUGEDA, MD, Principal Investigator — HOSPITAL UNIVERSITARIO INFANTA SOFIA; SILVIA CALDES, MD, Study Chair — HOSPITAL UNIVERSITARIO INFANTA SOFIA; YESIKA AMEZQUITA, MD, Study Chair — CLINICA FUENSANTA; JUAN MANUEL LOPEZ, PhD, Study Chair — HOSPITAL UNIVERSITARIO GREGORIO MARAÑON; SORAYA ABAD, MD, Study Chair — HOSPITAL UNIVERSITARIO GREGORIO MARAÑON; INES ARAGONCILLO, MD, Study Chair — Hospital Infanta Sofia; BORJA QUIROGA, MD, Study Chair — HOSPITAL GREGORIO MARAÑON; FERNANDO DE ALVARO, PhD, Study Chair — Hospital Infanta Sofia
Locations (5):
- Spain (5):
  - Hospital Universitario Infanta Sofia, San Sebastián de los Reyes, Madrid
  - Centro de Diálisis Los Enebros, Madrid
  - Hospital Universitario Gregorio Marañon, Madrid
  - Dialcentro, Madrid
  - Clinica Fuensanta, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aragoncillo I, Abad S, Caldes S, Amezquita Y, Vega A, Cirugeda A, Moratilla C, Ibeas J, Roca-Tey R, Fernandez C, Macias N, Quiroga B, Blanco A, Villaverde M, Ruiz C, Martin B, Ruiz AM, Ampuero J, de Alvaro F, Lopez-Gomez JM. Adding access blood flow surveillance reduces thrombosis and improves arteriovenous fistula patency: a randomized controlled trial. J Vasc Access. 2017 Jul 14;18(4):352-358. doi: 10.5301/jva.5000700. Epub 2017 Apr 20. PMID 28430315
- [Derived] Aragoncillo I, Amezquita Y, Caldes S, Abad S, Vega A, Cirugeda A, Moratilla C, Ibeas J, Roca-Tey R, Fernandez C, Quiroga B, Blanco A, Villaverde M, Ruiz C, Martin B, Ruiz AM, Ampuero J, Lopez-Gomez JM, de Alvaro F. The impact of access blood flow surveillance on reduction of thrombosis in native arteriovenous fistula: a randomized clinical trial. J Vasc Access. 2016 Jan-Feb;17(1):13-9. doi: 10.5301/jva.5000461. Epub 2015 Sep 18. PMID 26391583